CLINICAL TRIAL: NCT05312970
Title: A Phase 4 Randomized Trial Comparing Varithena to Endothermal Ablation for the Treatment of the Great Saphenous Vein
Brief Title: Varithena Versus Endothermal Ablation of the Great Saphenous Vein (VERITAS)
Acronym: VERITAS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment challenges and a difficult insurance coverage landscape
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S2473
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Varicose Veins
Keywords: Great Saphenous Vein Incompetence
MeSH Terms: conditions — Varicose Veins | interventions — Polidocanol; Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial 1:1 assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Varithena® (Active Comparator): Varithena® (polidocanol injectable foam) 1%
  Interventions: Drug: Varithena®
- FDA-approved ETA systems (Active Comparator): FDA-approved ETA systems, including Radiofrequency ablation (RFA) systems or Endovenous laser ablation (EVLA) systems.
  Interventions: Device: FDA-approved Endothermal Ablation (ETA) systems

INTERVENTIONS:
Drug: Varithena® — Varithena® (polidocanol injectable foam) 1%
  Arms: Varithena®
Device: FDA-approved Endothermal Ablation (ETA) systems — FDA-approved ETA systems, including Radiofrequency ablation (RFA) systems or Endovenous laser ablation (EVLA) systems.
  Arms: FDA-approved ETA systems

SUMMARY:
The purpose of this study is to observe insights into the benefits of Varithena compared to Endothermal Ablation (ETA) in the treatment of the great saphenous vein.

DETAILED DESCRIPTION:
To collect comparative evidence on patient reported outcomes of Varithena compared to ETA when used to treat the incompetent great saphenous vein (GSV). ETA will include either radiofrequency ablation or endovenous laser ablation according to the site's standard practice. To provide long term (1-year, 2-year, and 3-year) outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Primary GSV incompetence, defined as reflux > 0.5 seconds on Duplex ultrasound in a single limb (Note the contralateral limb can have varicosities or SVI if intervention is not required within 3 months i.e. asymptomatic)
* Failed conservative therapy (compression, diet, exercise, leg elevation)
* CEAP Clinical Condition Classification C2 - C6
* Vein diameter 5-10mm, inclusive
* GSV treatable length > 10cm
* Superficial venous disease manifest by clinical symptoms (rVCSS ≥ 4)
* Able to comprehend and sign an informed consent document and complete written study questionnaires
* Willing and able to return for scheduled follow-up visits (7-days, 3-months, 6-months, 12-months, 24-months, and 36-months post-procedure)
* Willingness to comply with post-treatment compression protocol

Exclusion Criteria:

* Allergy to polidocanol, xylocaine, or epinephrine
* Deep vein thrombosis or pulmonary embolism within 3 months prior to randomization or hypercoagulable disorder
* Post thrombotic deep vein disease above the calf veins
* Pregnancy or lactating (within 30 days of randomization)
* Symptomatic peripheral arterial disease or ankle-brachial pressure index (ABPI) < 0.8
* Previous treatment to targeted incompetent GSV or previous superficial thrombophlebitis in targeted GSV
* Previous venous intervention in affected limb in past 3 months
* Local aneurysmal GSV segments
* Inability to walk unaided
* Inability to wear post-procedure compression bandaging and stockings
* Patients with clinically significant reflux of the small saphenous vein (SSV) or anterior accessory saphenous vein (AASV)
* In the clinical judgement of the investigator, patient who will require ipsilateral deep venous intervention within 3 months following randomized treatment
* In the clinical judgement of the investigator, patient who will require contralateral venous intervention (superficial or deep) within 3 months following randomized treatment
* Patient on therapeutic anticoagulants
* Active malignancy
* Life expectancy < 2 years
* Documented COVID-19 infection currently or within 2 months prior to randomization
* Enrollment in another clinical trial that could confound the endpoint within 3 months prior to screening or within 3 months following enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Change in Varicose Veins Symptoms Questionnaire (VVSymQ) | Baseline to 3-month post treatment
  Mean change in Varicose Veins Symptoms Questionnaire (VVSymQ) between baseline and 3-month post treatment

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Vascular Care Connecticut, Darien, Connecticut
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Vein Healthcare Center, South Portland, Maine
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Columbia University Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - UT Physicians Cardiothoracic and Vascular Surgery, Houston, Texas
  - Lake Washington Vascular, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No